CLINICAL TRIAL: NCT06501651
Title: A Prospective, Randomized, Controlled, Multicenter Study of Sacubitril/Valsartan in the Treatment of Patients With Mild to Moderate Essential Hypertension and Type 2 Diabetic Nephropathy: The Hyper-Save Study
Brief Title: Sacubitril/Valsartan Treats Patients With Essential Hypertension and Type 2 Diabetic Nephropathy
Acronym: Hyper-Save
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Collaborators: The Second Affiliated Hospital of Chongqing Medical University (Other); Nanchong Central Hospital (Other Government); The People's Hospital of Leshan (Other); The Affiliated Traditional Chinese Medicine Hospital Of Southwest Medical University (Unknown); Chengdu First People's Hospital (Other); Mianyang People's Hospital (Unknown); Guan'an People's Hospital (Unknown); Meishan Traditional Chinese Medicine Hospital (Other); Qijiang District People's Hospital (Unknown); Meishan People's Hospital (Unknown); The First People's Hospital of Guangyuan (Unknown); Dazhou Central Hospital (Other)
Responsible Party: Principal Investigator, tianwenjie1976, Chief Physician, Sichuan Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ethical Review 2024(15-1)
Record Dates: First submitted 2024-06-28; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Essential Hypertension; Type 2 Diabetes; Nephropathy
Keywords: Essential hypertension; Type 2 diabetes; Nephropathy; Sacubitril/Valsartan
MeSH Terms: conditions — Essential Hypertension; Diabetes Mellitus, Type 2; Kidney Diseases | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Controlled, Multicenter Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Initial Dose: The starting dose of Sacubitril/Valsartan is 200 mg once daily. Dose Adjustment: If blood pressure targets (SBP < 130 mmHg and DBP < 80 mmHg) are not achieved after 2 weeks of treatment, the dose of Sacubitril/Valsartan should be doubled to 400 mg once daily.
  Additional Treatment: If blood pressure targets are still not met after an additional 2 weeks of treatment, Nifedipine controlled-release tablets (30 mg once daily) should be added to the regimen.
  Interventions: Drug: Sacubitril/Valsartan
- Comparator (Active Comparator): Initial Dose: The starting dose of Valsartan is 80 mg once daily. Dose Adjustment: If blood pressure targets (SBP < 130 mmHg and DBP < 80 mmHg) are not achieved after 2 weeks of treatment, the dose of Valsartan should be doubled to 160 mg once daily.
  Additional Treatment: If blood pressure targets are still not met after an additional 2 weeks of treatment, Nifedipine controlled-release tablets (30 mg once daily) should be added to the regimen.
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril/Valsartan — Sacubitril/Valsartan is a novel antihypertensive medication composed of an angiotensin II receptor blocker (ARB) Valsartan and a neprilysin inhibitor Sacubitril in a 1:1 molar co-crystal form. Sacubitril is a prodrug that, once ingested, is metabolized by esterases into its active form, which inhibits neprilysin activity. Neprilysin has various substrates, including natriuretic peptides and angiotensin II (Ang II). By inhibiting neprilysin, the levels of natriuretic peptides that have antihypertensive and organ-protective effects are increased. The other component, Valsartan, effectively inhibits the Ang II type 1 receptor (AT1R), providing additional antihypertensive and organ-protective effects. The co-crystal structure ensures that Sacubitril and Valsartan have similar absorption and elimination rates, thereby synchronizing their pharmacological effects.
  Arms: Experimental
Drug: Valsartan — Valsartan, effectively inhibits the Ang II type 1 receptor (AT1R), providing both antihypertensive and organ-protective effects.
  Arms: Comparator

SUMMARY:
This study aims to compare the efficacy and safety of Sacubitril/Valsartan versus Valsartan in patients with essential hypertension and type 2 diabetic nephropathy over a 12-week treatment period, including two treatment groups, with a total of 297 eligible subjects randomly assigned in a 2:1 ratio to either the experimental group or the control group.Subjects will participate in the study through two phases: the screening period and the follow-up period.The primary outcome measure is the change in systolic blood pressure from baseline after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, no gender restriction;
* Diagnosed with mild to moderate primary hypertension (140 ≤ SBP < 180 mmHg and/or 90 ≤ DBP < 110 mmHg), including newly diagnosed or inadequately treated patients (those who have not followed previous medical advice and have uncontrolled blood pressure according to the investigator);
* Diagnosed with type 2 diabetes (according to Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition)), and meeting the following conditions: a) Continuously on ≥ 1 glucose control medication regimens (which may include long-acting insulin) for at least 12 weeks before screening, with a stable treatment regimen (i.e., the same medication and dosage) for at least 28 days before screening, and maintaining this regimen during the study. At the investigator's discretion, the dose of supplemental short-acting insulin can be adjusted as needed to achieve adequate glucose control; b) HbA1c level ≤ 10.5% and fasting (≥ 8 hours) plasma glucose level ≤ 13.3 mmol/L (if fasting glucose > 13.3 mmol/L, the investigator may repeat the test to determine eligibility);
* Urine albumin/creatinine ratio (UACR) ≥ 30 mg/g in two measurements taken on separate days or eGFR < 60 mL/min/1.73 m²;
* Non-pregnant or fertile patients (male or female) using reliable contraception;
* Female patients with potential for pregnancy must have a negative pregnancy test at screening;
* Subjects must voluntarily agree to comply strictly with the study protocol requirements and sign a written informed consent form.

Exclusion Criteria:

* Presence of severe hypertension, malignant hypertension, hypertensive emergencies, or hypertensive crises;
* History or evidence of secondary hypertension within 12 months before screening, including but not limited to any of the following: renovascular hypertension, renal parenchymal hypertension, unilateral or bilateral renal artery stenosis, coarctation of the aorta, primary aldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, and drug-induced hypertension;
* History of angioedema (drug-related or other causes) within 12 months before screening;
* Presence of diabetic ketoacidosis;
* History or evidence of secondary diabetes within 12 months before screening, including but not limited to any of the following: endocrine disorders causing carbohydrate metabolism disorders, pancreatogenic diabetes, hepatogenic diabetes, nephrogenic diabetes, etc.;
* History of malignancy in any organ system (excluding localized basal cell carcinoma of the skin);
* History of acute stroke, lacunar infarction, or dementia within 6 months before screening;
* History of coronary artery bypass graft surgery or any percutaneous coronary intervention (PCI) within 6 months before screening;
* Previously diagnosed or currently diagnosed heart failure (NYHA Class III-IV) or clinically significant valvular heart disease;
* History or current diagnosis of cardiac abnormalities: (1) second or third-degree atrioventricular block without a pacemaker; (2) clinically significant arrhythmias, including atrial fibrillation with a ventricular rate ≥ 120 bpm; (3) family history of long QT syndrome or torsades de pointes ventricular tachycardia;
* Chronic kidney disease stage 4 or higher (eGFR < 30 mL/min/1.73 m²), receiving renal dialysis, or history of kidney transplantation;
* Significant abnormalities in laboratory tests, such as potassium levels > 5.5 mmol/L or < 3.5 mmol/L, sodium levels < 130 mmol/L, liver function (ALT, AST) results > 3 times the upper limit of normal;
* History of allergy to antihypertensive drugs such as ARBs, Angiotensin-Converting Enzyme (ACE) inhibitors, or renin inhibitors;
* Clear history of intolerance to drugs similar to the study medication (e.g., ACE inhibitors, ARBs);
* Use of traditional Chinese or Western medicines that could affect the study's efficacy during the study period (see appendix for list);
* Any surgery or medical condition that significantly alters the absorption, distribution, metabolism, or excretion of any medication, including but not limited to the following: clinically significant gastrointestinal surgery within 12 months before the screening (e.g., gastrectomy, gastrointestinal anastomosis, bowel resection, gastric bypass, gastroenterostomy, or gastric banding), current active inflammatory bowel disease or history of active inflammatory bowel disease;
* Pregnant or breastfeeding women, or patients of childbearing potential unwilling or unable to use effective contraception during the study period;
* Participation in another clinical study using any investigational drug or observational study within 30 days before screening;
* Other conditions that, in the investigator's judgment, may affect the conduct of the clinical study or the determination of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Reduction in 24-hour ambulatory systolic blood pressure(SBP) | From enrollment to the end of treatment at 12 weeks
  The comparison of the reduction in 24-hour ambulatory systolic blood pressure from baseline between the two groups

SECONDARY OUTCOMES:
Reduction in 24-hour ambulatory diastolic blood pressure(DBP) | From enrollment to the end of treatment at 12 weeks
  The comparison of the reduction in 24-hour ambulatory diastolic blood pressure from baseline between the two groups
Changes in daytime and nighttime ambulatory blood pressure | From enrollment to the end of treatment at 12 weeks
  The comparison of the changes in daytime and nighttime ambulatory blood pressure between the two groups. (The mean daytime blood pressure is defined as the average of hourly measurements taken between 6:00 and 22:00, and the mean nighttime is defined as the average of hourly measurements taken between 22:00 and 6:00.)
Rate of dipper blood pressure restoration | From enrollment to the end of treatment at 12 weeks
  The comparison of the proportion of subjects in each group who achieve a dipper blood pressure pattern, defined as a nighttime blood pressure reduction of 10-20% in both systolic and diastolic blood pressure.
Rate of blood pressure achievement | From enrollment to the end of treatment at 12 weeks
  The comparison of the proportion of subjects in each group who achieve blood pressure targets (SBP < 130 mmHg and DBP < 80 mmHg)
Rate of hypertension treatment response | From enrollment to the end of treatment at 12 weeks
  The comparison of the proportion of subjects in each group who achieve hypertension treatment response, defined as: SBP < 140 mmHg and/or a reduction from baseline of ≥ 20 mmHg; DBP < 90 mmHg and/or a reduction from baseline of ≥ 10 mmHg; both of them
Improvement in diabetes condition | From enrollment to the end of treatment at 12 weeks
  Comparison of reductions in fasting plasma glucose (FPG) and glycated hemoglobin (HbA1c) between the two groups
Improvement in Renal Function | From enrollment to the end of treatment at 12 weeks
  The comparison of reductions in serum creatinine, urine albumin/creatinine ratio, and blood urea nitrogen between the two groups
Medication utilization | From enrollment to the end of treatment at 12 weeks
  The comparison of dose escalation proportions and the proportion of subjects requiring adjunctive nifedipine controlled-release tablets between the two groups
Safety assessments | From enrollment to the end of treatment at 12 weeks
  Safety assessments included monitoring of all adverse events (AEs), serious AEs (SAEs), and regular monitoring of vital signs and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Academy of Medical Sciences · Sichuan Provincial People's Hospital, Chengdu, Sichuan, China